CLINICAL TRIAL: NCT02402387
Title: The Influence of Head and Neck Position on the Oropharyngeal Leak Pressure Using Air-Q SP Airway
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Diagnostic
Other Study IDs: 4-2015-0050
Record Dates: First submitted 2015-03-24; First posted 2015-03-30 (Estimated); Last update posted 2017-01-25 (Estimated); Status verified 2017-01

CONDITIONS: General Anesthesia

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Neutral (Active Comparator): The patient's head will be in neutral position.
  Interventions: Procedure: Neutral head position; Device: Air-Q SP Airway
- Flexed (Experimental): The patient's head will be flexed.
  Interventions: Procedure: Flexed head position; Device: Air-Q SP Airway
- Extended (Experimental): The patient's head will be extended.
  Interventions: Procedure: Extended head position; Device: Air-Q SP Airway
- Rotated (Experimental): The patient's head will be rotated.
  Interventions: Procedure: Rotated head position; Device: Air-Q SP Airway

INTERVENTIONS:
Procedure: Neutral head position
  Arms: Neutral
Procedure: Flexed head position
  Arms: Flexed
Procedure: Extended head position
  Arms: Extended
Procedure: Rotated head position
  Arms: Rotated
Device: Air-Q SP Airway

SUMMARY:
The purpose of this study is to investigate the changes of the oropharyngeal leak pressure of the air-Q self-pressurizing masked laryngeal airway in the different head and neck positions. Moreover, the adequacy of ventilation will be assessed in the different head and neck positions.

ELIGIBILITY:
Inclusion Criteria:

* adult patients aged over 20 yrs who are scheduled for surgery under general anesthesia

Exclusion Criteria:

* anticipated difficult intubation
* body mass index more than 30 km/m2
* history of gastroesophageal reflux disease
* history of esophageal operation
* cervical spine disease
* mass in the oral cavity or neck

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2015-05-12 (Actual); Primary Completion 2015-08-27 (Actual); Study Completion 2015-08-27 (Actual)

PRIMARY OUTCOMES:
Oropharyngeal leak pressure | Within 5 minutes after the insertion of the air-q self-pressurizing masked laryngeal airway
  The oropharyngeal leak pressure was measured by closing the expiratory valve of the circle system at fixed O2 flow 3L/min and 40 cmH2O

SECONDARY OUTCOMES:
Peak airway pressure | Within 5 minutes after the insertion of the air-q self-pressurizing masked laryngeal airway
Fiberoptic bronchoscope grade | Within 5 minutes after the insertion of the air-q self-pressurizing masked laryngeal airway

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Anesthesiology and Pain Medicine, Yonsei University College of Medicine, Seoul, Seoul, South Korea

REFERENCES:
- [Derived] Kim HJ, Lee K, Bai S, Kim MH, Oh E, Yoo YC. Influence of head and neck position on ventilation using the air-Q(R) SP airway in anaesthetized paralysed patients: a prospective randomized crossover study. Br J Anaesth. 2017 Mar 1;118(3):452-457. doi: 10.1093/bja/aew448. PMID 28203730